CLINICAL TRIAL: NCT04093037
Title: Analysis of the Diagnostic Performance of LacryDiag, a New "All-in-one" Non-contact Analyzer of the Ocular Surface in the Dry Eye. Study LACRYMOSA
Brief Title: Analysis of the Diagnostic Performance of LacryDiag, a New Analyzer of the Ocular Surface in the Dry Eye
Acronym: LACRYMOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18CH115; 2018-A02257-48 (Other: ANSM)
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye
Keywords: Dry eye; LacryDiag; Fluorescein; Break-Up Time (BUT); Schirmer test; Lacrimal film; Oxford score; Meibomian Gland; Tear Meniscus (TM); Non Invasive Break-Up Time (NIBUT)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: 80 patients divided into 4 subgroups according to the value of manual Standard Break-Up-Time (SBUT):
  * 0-5 seconds (very dry)
  * 5-10 seconds (sec)
  * 10-15 seconds (moderately dry)
  * 15-20 seconds (normal)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with dry eye disease (Experimental): Patient with dry eye disease will be included. They will have:
  * Time #1: LacryDiag examination without dye
  * Time #2: MicroInstillation Break-Up Time (MIBUT) + Oxford score
  * Time #3: Standard Break-Up Time (SBUT)
  * Time #4: Schirmer test
  * Satisfaction questionnaire to the patient
  Interventions: Diagnostic Test: Time #1: Non Invasive Break-Up Time (NIBUT); Diagnostic Test: Time #2: MicroInstillation Break-Up Time (MIBUT) + Oxford score; Diagnostic Test: Time #3: Standard Break-Up Time (SBUT); Diagnostic Test: Time #4: Schirmer test; Diagnostic Test: Satisfaction questionnaire to the patient

INTERVENTIONS:
Diagnostic Test: Time #1: Non Invasive Break-Up Time (NIBUT) — A LacryDiag examination without dye will be realized. All measurements are made without contact. It's calculates the Non Invasive Break-Up Time (NIBUT), Tear Meniscus (TM) height (in millimeters) and number of Meibomian Gland.
  These are different pictures taken with LacryDiag and analyzed.
  Other Names: LacryDiag; Complete diagnosis of dry eyes
Diagnostic Test: Time #2: MicroInstillation Break-Up Time (MIBUT) + Oxford score — The MicroInstillation of fluorescein Break-Up Time (MIBUT) will be calculated by manual MIBUT and LacryDiag MIBUT.
  The Oxford score will be calculated. It's used to clinically determine the severity of dry eyes with minimum score at 0 (none) and maximum score at 5 (very severity).
Diagnostic Test: Time #3: Standard Break-Up Time (SBUT) — The Standard Break-Up Time (SBUT) with fluorescein macroinstillation will be calculated by manual SBUT and LacryDiag SBUT.
Diagnostic Test: Time #4: Schirmer test — The Schirmer test will be performed. It consists of applying the end of a small strip of blotting paper behind the lower eyelid and examining the strip after 5 minutes.
Diagnostic Test: Satisfaction questionnaire to the patient — A satisfaction questionnaire to the patient will be completed at the end of the participation at the study.

SUMMARY:
LacryDiag is a new Conformity European (CE) marked diagnostic imaging device devoted to the analysis of the ocular surface. It is an "all in one" device that provides 4 data: non-invasive break-up time (Non-Invasive Break-Up-Time (NIBUT) without fluorescein eye drop); height of the Tear Meniscus (TM); an infrared image of the meibomian glands; a picture of the lacrimal film by interferometry. it's performance will be compare between in diagnosing dry eye syndrome with the standard clinical evaluation, in 80 patients suffering from dry eye diseases and followed at the consultation of the Ophthalmology department of the University Hospital of Saint-Etienne.

DETAILED DESCRIPTION:
The primary purpose of this study is to compare the value of Break-Up-Time (BUT) between Non-Invasive Break-Up-Time (NIBUT) measured by LacryDiag and Standard Break-Up-Time (SBUT) measured by usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Affiliates or beneficiaries of social security scheme
* With Dry eye of any cause, diagnosed with conventional means
* Signed informed consent

Exclusion Criteria:

* Major blepharospasm
* Serious illness preventing participation according to investigator
* Allergy to fluorescein
* Pregnant or / and breastfeeding women
* Under guardianship, curatorship or safeguard of justice
* Unable to express their consent
* Person in emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Break-Up-Time (BUT) | Day: 1
  Comparison of Break-Up-Time (BUT) measured by 2 methods : LacryDiag Non Invasive Break-Up Time (NIBUT) and manual Standard Break-Up Time (SBUT).
  Measured in seconds by time#1: Non Invasive Break-Up Time (NIBUT) and time#3: Standard Break-Up Time (SBUT).

SECONDARY OUTCOMES:
Standard Break-Up Time (SBUT) | Day: 1
  Comparison of Standard Break-Up Time (SBUT) between LacryDiag SBUT results and manual SBUT results. Measured in seconds.
  Measured by time#3: Standard Break-Up Time (SBUT).
MicroInstillation Break-Up Time (MIBUT) | Day: 1
  Comparison of MicroInstillation Break-Up Time (MIBUT) between LacryDiag MIBUT results and manual MIBUT results.
  Measured in seconds by time#1: Non Invasive Break-Up Time (NIBUT) and time#2: MicroInstillation Break-Up Time (MIBUT).
Tear Meniscus (TM) height and Schirmer test | Day: 1
  Correlation between Tear Meniscus (TM) height (in millimeters) and Schirmer test (in millimeters).
  Measured by time#1: Non Invasive Break-Up Time (NIBUT) and time#4: Schirmer test.
Percentage loss of Meibomian Gland. | Day: 1
  Measured by time#1: Non Invasive Break-Up Time (NIBUT).
Thickness (in nanometer) and regularity of lacrimal film (type) | Day: 1
  Correlation between measure thickness (in nanometer) and regularity of lacrimal film (type).
  Measured by time#1: Non Invasive Break-Up Time (NIBUT).

CONTACTS AND LOCATIONS:
Overall Officials: Gilles THURET, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No